CLINICAL TRIAL: NCT04257708
Title: Cavity Evaluation Before Intracytoplasmic Sperm Injection in Women With Infertility
Brief Title: Cavity Evaluation Before Intracytoplasmic Sperm Injection
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Aljazeera Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Uterus
Record Dates: First submitted 2020-02-04; First posted 2020-02-06 (Actual); Last update posted 2020-02-06 (Actual); Status verified 2020-02

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- normal uterine cavity
  Interventions: Diagnostic Test: ultrasound
- abnormal uterine cavity
  Interventions: Diagnostic Test: ultrasound

INTERVENTIONS:
Diagnostic Test: ultrasound — Transvaginal us to assess the cavity

SUMMARY:
Uterine cavity evaluation is an integral part of assessment Of women for ICSI

DETAILED DESCRIPTION:
Transvaginal us is the main role in this aspect

ELIGIBILITY:
Inclusion Criteria:

* women with infertility more than one year

Exclusion Criteria:

* 2omen with medical disorders

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Infertile women
Study Population: Women with infertility
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-02-09 (Estimated); Primary Completion 2020-11-10 (Estimated); Study Completion 2021-01-10 (Estimated)

PRIMARY OUTCOMES:
The number of women who will has positive pregnancy test | within a year
  The women who will got pregnant

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud Alalfy, PhD, Study Chair — Algezeera
Locations (1):
- Algazeerah, Giza, Egypt